CLINICAL TRIAL: NCT04870242
Title: Enhanced Recovery After Surgery in Pediatric Surgery in Jordan: A Retrospective Cohort Study in a Tertiary University Hospital
Brief Title: Studding the Implementation of ERAS Protocols in Pediatric Surgery
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Ahmad Abu-Shanab, Dr., University of Jordan
Other Study IDs: 67/2019/6216
Record Dates: First submitted 2021-04-29; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: ERAS; Pediatric Disorder; Appendicitis; Hydrocele
Keywords: Enhanced recovery after surgery (ERAS); enhanced recovery protocol; fast-track surgery; pediatric surgery
MeSH Terms: conditions — Appendicitis; Testicular Hydrocele | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pediatric surgery patients: all pediatric surgery patients, aged from 6 months up to 18 years, underwent surgery between January 2017 to December 2018
  Interventions: Other: Observational study, non-interventional

INTERVENTIONS:
Other: Observational study, non-interventional — observational study for the ERAS protocols in pediatric surgery

SUMMARY:
this is a retrospective cohort, descriptive study, investigating the role of ERAS protocols, in pediatric surgery and evaluate the feasibility and effectiveness of implementing these protocols

ELIGIBILITY:
Inclusion Criteria:

* all patients aged 6months -18 years, who underwent pediatric surgeries at a single tertiary institution

Exclusion Criteria:

* patients who had co-morbidities that might affect the outcome of the enhanced recovery and those who were younger than 6 months.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: all patients aged 6months -18 years, who underwent pediatric surgeries at a single tertiary institution
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Duration of Hospital stay, | retrospectively studied. data collection done at least 1 year after surgery
Total Hospital expenses | retrospectively studied. data collection done at least 1 year after surgery
readmission within 30 days | retrospectively studied. data collection done at least 1 year after surgery
reoperation within 90 days | retrospectively studied. data collection done at least 1 year after surgery
post op ER visits | retrospectively studied. data collection done at least 1 year after surgery
Pain control, according to a scale from 0-10, post-operative pain after implementation of ERAS protocols | retrospectively studied. data collection done at least 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Raed Al-Taher, M.D, Principal Investigator — University of Jordan
Locations (1):
- University Of Jordan, Amman, Amman, Jordan, Jordan

IPD SHARING:
Plan to Share IPD: No